CLINICAL TRIAL: NCT04098198
Title: Biomarkers for Inborn Errors of Metabolism: An International, Multicenter, Observational, Longitudinal Protocol
Brief Title: Biomarkers for Inborn Errors of Metabolism
Acronym: BioMetabol
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BioMetabol
Record Dates: First submitted 2019-08-23; First posted 2019-09-23 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2021-05

CONDITIONS: Inborn Errors of Metabolism; Biomarker
Keywords: Inborn Error of Metabolism; Biomarker
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with an Inborn Error of Metabolism: Participants diagnosed with an Inborn Error of Metabolism aged between 2 months to 50 years

SUMMARY:
International, multicenter, observational, longitudinal study to identify or monitor Inborn Error of Metabolism disease biomarkers and to explore the clinical robustness, specificity, and long-term variability of these biomarkers

DETAILED DESCRIPTION:
Inborn Errors of Metabolism (IEM) are a large group of congenital metabolic disorders, resulting from the absence or abnormality of an enzyme or its cofactor and leading to either accumulation or deficiency of a specific metabolite. More than 800 IEM have been described in the literature, with a widely accepted classification focusing on the main substrate which is affected.

Clinical phenotypes of IEM are broad and often non-specific, mimicking more common conditions, and the onset of symptoms can occur at any age, from fetus to adult. Peroxisomal and lysosomal storage disorders, for example, often have characteristic clinical features and permanent, progressive symptoms that are independent of triggering events (e.g. anemia, thrombocytopenia, and hepatomegaly in a child of Ashkenazi-Jewish ancestry is suggestive of Gaucher disease) 6. More common findings include hypoketotic hypoglycemia, lactic acidosis, metabolic acidosis, ketosis, hyperammonemia, or other metabolic acidosis in combination with hyperammonemia.

The goal of treatment for participants with IEM are the prevention of further accumulation of harmful substances, correction of metabolic abnormalities, and elimination of toxic metabolites. Most participants suffering for rare metabolic diseases start with very severe phenotypes and with rapid progression of the disease that often leads to irreversible damage of their organs. A quick diagnosis is necessary for urgent treatment.

Biomarkers serve as measurable indicators of normal biological or pathological processes. They are typically directly linked to genetic variants in specific genes and can predict, diagnose, monitor and assess the severity of a disease.

CENTOGENE has an outstanding experience regarding the investigation and development of biomarkers for IEM. Given the large amount of participants CENTOGENE is facing and diagnosing, it has a big repertoire of samples to use for the biomarker characterization. This led for example to the identification of Lyso-Gb1 as a novel biomarker for Gaucher disease orLyso-SM509 for Niemann-Pick Disease. The established workflows and gained knowledge for the biomarker development at CENTOGENE will enhance the search for new biomarkers of other IEM.

It is the goal of this study to identify, validate, and monitor biochemical markers from affected participants for Inborn Errors of Metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant or from their parent/legal guardian, before any study related procedures
* The participant aged between 2 months old and 50 years old
* The diagnosis of an Inborn Error of Metabolism is genetically confirmed

Exclusion Criteria:

* Inability to provide informed consent
* The participant is younger than 2 months old or older than 50 years old
* The diagnosis of an Inborn Error of Metabolism (IEM) is not genetically confirmed
* Previously enrolled in the study

Ages: 2 Months to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants with an Inborn Error of Metabolism
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Identification of biomarkers for Inborn Errors of Metabolism | 2 years
  All samples will be analyzed for the identification of biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

SECONDARY OUTCOMES:
Exploring the clinical robustness, specificity, and long-term variability of biomarkers for Inborn Errors of Metabolism | 2 years
  Samples will be analyzed for the identified biomarker candidates via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof. Dr., Study Chair — Centogene GmbH
Locations (13):
- University Hospital Center Mother Teresa, Tirana, Albania
- Egypt (6):
  - Department of Clinical Genetics, Alexandria University Children's Hospital, Alexandria
  - Department of Pediatrics, Alexandria University Children's Hospital, Alexandria
  - Department of Medical Genetics ,Faculty of Medicine, Ain Shams University, Cairo
  - Ain Shams University, Cairo
  - Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo
  - Pediatrics Departmnet, Tanta University, Tanta
- Department of Molecular and Medical Genetics , Tbilisi State Medical University, Tbilisi, Georgia
- Amrita Institute of Medical Sciences, Kerola, India
- Children's hospital, Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania
- Departmnet of Pediatric Gastroenterology and Hepatology, The Children's Hospital and Institute of Child Health, Lahore, Pakistan
- Emergency Hospital for Children "Louis Turcanu", Timișoara, Romania
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CENTOGENE is a rare disease company focused on transforming clinical, genetic, and biochemical data into medical solutions for Patients — https://www.centogene.com/